CLINICAL TRIAL: NCT00219284
Title: A Prospective, Multi-center, Randomized, Open-label Study With Blinded Raters to Evaluate the Effects of Immediate Versus Delayed Switch to Carbidopa/Levodopa/Entacapone on Motor Function and Quality of Life in Patients With Parkinson's Disease With End-of-dose Wearing Off
Brief Title: Effects of Carbidopa/Levodopa/Entacapone on Motor Function and Quality of Life in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CELC200AUS11
Record Dates: First submitted 2005-06-30; First posted 2005-09-22 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease With End of Dose Wearing Off
Keywords: Parkinson's disease, tremor
MeSH Terms: conditions — Parkinson Disease; Tremor | interventions — Stalevo

ARMS (2):
- Immediate switch (Experimental): Patients were switched the day after randomization from combined carbidopa/levodopa to combined carbidopa/levodopa/entacapone. Patients received the same doses of carbidopa (12.5, 25.0, or 37.5 mg) and levodopa (50, 100, or 150 mg) they were receiving prior to the switch, combined with 200 mg of entacapone. The frequency of doses per day prior to the switch remained the same after the switch.
  Interventions: Drug: Carbidopa/levodopa/entacapone
- Delayed switch (Active Comparator): Patients were switched 4 weeks after randomization from combined carbidopa/levodopa to combined carbidopa/levodopa/entacapone. Patients received the same doses of carbidopa (12.5, 25.0, or 37.5 mg) and levodopa (50, 100, or 150 mg) they were receiving prior to the switch, combined with 200 mg of entacapone. The frequency of doses per day prior to the switch remained the same after the switch.
  Interventions: Drug: Carbidopa/levodopa/entacapone

INTERVENTIONS:
Drug: Carbidopa/levodopa/entacapone — Carbidopa/levodopa/entacapone was administered in 1 of 3 dose combinations: 12.5/50/200 mg, 25/100/200 mg, or 37.5/150/200 mg. The selected combination dose contained the same doses of carbidopa and levodopa the patient was receiving prior to switching to carbidopa/levodopa/entacapone.

SUMMARY:
To assess motor function and quality of life (QoL) in Parkinson's disease (PD) subjects with end-of-dose wearing off, comparing immediate and delayed switch to carbidopa/levodopa and entacapone.

DETAILED DESCRIPTION:
This was a prospective, multi-center, randomized, open-label study with blinded raters to evaluate the effects of immediate versus delayed switch to carbidopa/levodopa/entacapone on motor function and quality of life in patients with Parkinson's disease with end-of-dose wearing off.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 30-80 years of age (inclusive). Patients aged 81-85 years were eligible to participate if the principal investigator considered the patient to be in otherwise good health.
* Clinical diagnosis of Parkinson's disease exhibiting two of three symptoms (rigidity, resting tremor, bradykinesia).
* All patients were required to have end-of dose wearing off (EODWO, re-emergence of PD symptoms at the end of at least two daily doses of levodopa during waking hours).
* Taking regular doses of immediate release carbidopa/levodopa

Exclusion Criteria:

* Unstable Parkinson's Disease requiring booster doses or treatment with as needed dose regimens of levodopa
* Female subjects who are pregnant, trying to become pregnant or nursing an infant

Other protocol-defined inclusion/exclusion criteria applied to this study.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (41):
  - Phoenix, Arizona
  - Fullerton, California
  - Irvine, California
  - La Jolla, California
  - Los Angeles, California
  - Pasadena, California
  - Reseda, California
  - Stanford, California
  - Fort Collins, Colorado
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Bradenton, Florida
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Naples, Florida
  - Palm Beach, Florida
  - Plantation, Florida
  - Pompano Beach, Florida
  - Port Charlotte, Florida
  - Chicago, Illinois
  - Flossmoor, Illinois
  - Lenexa, Kansas
  - Topeka, Kansas
  - Baltimore, Maryland
  - Bingham Farms, Michigan
  - Southfield, Michigan
  - Hattiesburg, Mississippi
  - Columbia, Missouri
  - St Louis, Missouri
  - Ridgewood, New Jersey
  - Commack, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Bellevue, Ohio
  - Canton, Ohio
  - Tualatin, Oregon
  - East Stroudsburg, Pennsylvania
  - Houston, Texas
  - Spokane, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Caroline, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Switch: Carbidopa/levodopa/entacapone was administered in 1 of 3 dose combinations: 12.5/50/200 mg, 25/100/200 mg, or 37.5/150/200 mg. The selected combination dose contained the same doses of carbidopa and levodopa the patient was receiving prior to switching to carbidopa/levodopa/entacapone. Patients were switched the day after randomization from combined carbidopa/levodopa to combined carbidopa/levodopa/entacapone. Patients received the same doses of carbidopa (12.5, 25.0, or 37.5 mg) and levodopa (50, 100, or 150 mg) they were receiving prior to the switch, combined with 200 mg of entacapone. The frequency of doses per day prior to the switch remained the same after the switch.
- Delayed Switch: Carbidopa/levodopa/entacapone was administered in 1 of 3 dose combinations: 12.5/50/200 mg, 25/100/200 mg, or 37.5/150/200 mg. The selected combination dose contained the same doses of carbidopa and levodopa the patient was receiving prior to switching to carbidopa/levodopa/entacapone. Patients were switched 4 weeks after randomization from combined carbidopa/levodopa to combined carbidopa/levodopa/entacapone. Patients received the same doses of carbidopa (12.5, 25.0, or 37.5 mg) and levodopa (50, 100, or 150 mg) they were receiving prior to the switch, combined with 200 mg of entacapone. The frequency of doses per day prior to the switch remained the same after the switch.
Period: Treatment Phase - 16 Weeks
Arm/Group | Immediate Switch | Delayed Switch
Started | 180 | 179
Completed | 136 | 128
Not Completed | 44 | 51
Not completed — Adverse Event | 26 | 24
Not completed — Abnormal laboratory value(s) | 0 | 1
Not completed — Lack of Efficacy | 3 | 10
Not completed — Protocol Violation | 9 | 5
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Lost to Follow-up | 1 | 2
Period: Extension Phase - 8 Weeks
Arm/Group | Immediate Switch | Delayed Switch
Started | 114 (Not all subjects who completed the treatment phase chose to enter this optional extension phase.) | 106 (Not all subjects who completed the treatment phase chose to enter this optional extension phase.)
Completed | 112 | 99
Not Completed | 2 | 7
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Switch | Delayed Switch | Total
Number analyzed (Participants) | 180 | 179 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.7 (9.18) | 68.3 (10.38) | 68.5 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 71 | 145
  Male | 106 | 108 | 214

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score From Baseline to Week 4
Description: Motor function was assessed with the UPDRS part III. There are 14 items in the instrument, each measured on a 5 point scale (0-4): Speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability, and body bradykinesia. The sum of scores can range from 0 to 56; a higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: Baseline to Week 4
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only patients with baseline and Week 4 UPDRS part III scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 161 | 167
Units on a scale | -3.7 (0.66) [-5.02 to -2.41] | -1.8 (0.58) [-2.95 to -0.68]

2. Secondary Outcome: Change in Parkinson's Disease Quality of Life Score From Baseline to Week 4
Description: Quality of life was assessed with the Parkinson's Disease Quality of Life Instrument (PDQUALIF), a 33-item self-reported questionnaire which includes seven domains: Social/role function, self-imaging/sexuality, sleep, outlook, physical function, independence, and urinary function. Questions are scored on a 5-point Likert scale ranging from 1 (never) to 3 (sometimes) to 5 (always). The 1 to 5 range was recoded to 0 to 4 for the analysis. The total score can range from 0 to 132. A lower score indicates better quality of life. A negative change score indicates improvement.
Time Frame: Baseline to Week 4
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only patients with baseline and Week 4 PDQUALIF scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 163 | 159
Units on a scale | -0.4 (0.88) [-4.51 to -0.53] | 1.1 (0.77) [-2.84 to 0.66]

3. Secondary Outcome: Change in Parkinson's Disease Quality of Life Score From Baseline to Week 8
Description: as for outcome 2
Time Frame: Baseline to Week 8
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only patients with baseline and Week 8 PDQUALIF scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 150 | 155
Units on a scale | -2.5 (1.01) | -1.1 (0.89)

4. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score From Baseline to Week 8
Description: Motor function was assessed with the UPDRS part III. There are 14 items in the instrument, each measured on a 5-point scale (0-4): Speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability, and body bradykinesia. The sum of scores can range from 0 to 56; a higher score indicates greater disability. A negative change score indicates improvement.
Time Frame: Baseline to Week 8
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only patients with baseline and Week 8 UPDRS part III scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 146 | 152
Units on a scale | -3.6 (0.71) | -3.7 (0.62)

5. Secondary Outcome: Change in the 39-item Parkinson's Disease Questionnaire (PDQ-39) Total Score From Baseline to Week 4
Description: The PDQ-39 is another instrument used to assess quality of life in individuals with Parkinson's disease. The questionnaire provides scores on eight scales: Mobility, activities of daily living, emotions, stigma, social support, cognition, communication, and bodily discomfort. Questions are scored on a 5-point Likert scale ranging from 1 (never) to 3 (sometimes) to 5 (always). The 1 to 5 range was recoded to 0 to 4 for the analysis. The total score can range from 0 to 156. A lower score indicates better quality of life. A negative change score indicates an improvement.
Time Frame: Baseline to Week 4
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only patients with baseline and Week 4 PDQ-39 scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 163 | 169
Units on a scale | -1.7 (1.34) | 0.8 (1.17)

6. Secondary Outcome: Change in the 39-item Parkinson's Disease Questionnaire (PDQ-39) Total Score From Baseline to Week 8
Description: as for outcome 5
Time Frame: Baseline to Week 8
Population: Intent-to-treat (ITT) population: All randomized patients who received at least one dose of study drug and had at least one post-baseline assessment of the primary efficacy variable. Only patients with baseline and Week 8 PDQ-39 scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 150 | 155
Units on a scale | -5.8 (1.48) | -1.9 (1.31)

7. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Score From Baseline to End of Treatment
Description: as for outcome 1
Time Frame: Baseline to end of treatment (Week 16 in the Immediate Switch group, Week 20 in the Delayed Switch group)
Population: ITT population - For each patient, the last post-baseline measurement during the treatment phase was used as the end-of-treatment measurement. Only patients with baseline and end-of-treatment UPDRS part III scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 176 | 171
Units on a scale | -3.6 (0.69) | -3.3 (0.64)

8. Secondary Outcome: Change in Parkinson's Disease Quality of Life Score From Baseline to End of Treatment
Description: as for outcome 2
Time Frame: Baseline to end of treatment (Week 16 in the Immediate Switch group, Week 20 in the Delayed Switch group)
Population: ITT population - For each patient, the last post-baseline measurement during the treatment phase was used as the end-of-treatment measurement. Only patients with baseline and end-of-treatment PDQUALIF scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 176 | 172
Units on a scale | -1.3 (0.97) | 0.2 (0.89)

9. Secondary Outcome: Change in the 39-item Parkinson's Disease Questionnaire (PDQ-39) Total Score From Baseline to End of Treatment
Description: as for outcome 5
Time Frame: Baseline to end of treatment (Week 16 in the Immediate Switch group, Week 20 in the Delayed Switch group)
Population: ITT population - For each patient, the last post-baseline measurement during the treatment phase was used as the end-of-treatment measurement. Only patients with baseline and end-of-treatment PDQ-39 scores were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 176 | 172
Units on a scale | -2.8 (1.60) | 0.4 (1.47)

ADVERSE EVENTS:
Arm/Group | Immediate Switch | Delayed Switch
Serious Adverse Events (participants affected / at risk) | 8/180 | 12/179
Other Adverse Events (participants affected / at risk) | 100/180 | 66/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Switch (N=180) | Delayed Switch (N=179)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Global amnesia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Switch (N=180) | Delayed Switch (N=179)
Constipation (Gastrointestinal disorders) | 10 | 6
Diarrhoea (Gastrointestinal disorders) | 29 | 21
Nausea (Gastrointestinal disorders) | 31 | 13
Fatigue (General disorders) | 12 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Dizziness (Nervous system disorders) | 16 | 13
Dyskinesia (Nervous system disorders) | 7 | 12
Tremor (Nervous system disorders) | 9 | 6
Depression (Psychiatric disorders) | 9 | 7
Chromaturia (Renal and urinary disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.